CLINICAL TRIAL: NCT00384800
Title: A Phase II Study of Tegafur/Uracil (UFUR®)Plus Thalidomide for the Treatment of Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-94037
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tegafur

INTERVENTIONS:
Drug: Thalidomide(THADO), Tegafur/Uracil(UFUR)

SUMMARY:
Primary objective:

To evaluate the overall response rate of tegafur/uracil (UFUR®) and thalidomide in the treatment of advanced or metastatic hepatocellular carcinoma.

Secondary objectives:

1. To determine the disease stabilization rate;
2. To assess the progression-free survival and overall survival;
3. To establish the safety profile;
4. To evaluate the changes of circulating factors indicating the angiogenesis activity and their correlation with objective tumor response.

DETAILED DESCRIPTION:
Thalidomide is a glutamic acid derivative first developed in 1950s, was marketed as a sedative, tranquilizer, and antiemetic for morning sickness.

It was withdrawn from the European and Canadian markets in early 1960s because of its teratogenic effects . It was not until 1998 when FDA approved thalidomide in the US for the treatment of erythema nodosum leprosum , ENL.

In recent years, thalidomide is emerging as a novel treatment for cancer because of its anti-angiogenic properties. The clinical efficacy has been demonstrated in various types of human cancers, such as myeloma, hormone-refractory prostate cancer, high-grade glioma, renal cell carcinoma, and melanoma.

UFUR® is a composite drug composed of 100mg tegafur and 224mg uracil (molar ratio:1:4). It was marketed as UFT® in Japan and marketed as UFUR® in Taiwan.

Tegafur, a prodrug of 5-FU, is easily absorbed though the gastro-intestinal tract slowly metabolized to 5-FU mainly in liver . Uracil is an inhibitor of dihydro-pyrimidine dehydrogenase (DPD), the rate-limiting enzyme of 5-FU degradation.

Tegafur/urail is expected to maintain a stably high concentration in liver and in circulation. Tegafur/uracil has been approved for the indications of advanced gastric cancer and colorectal cancer, which are traditionally indicated for the therapy of 5-FU-based chemotherapy, in Japan and Taiwan.

We hypothesize that combination of tegafur/uracil (UFUR®) and thalidomide, both of which have been shown to be active in some HCC patients, may be a highly useful regimen for the treatment of advanced HCC. There are several rationales underlying this combination. First, anti-angiogenesis therapy may improve the efficacy of chemotherapy by normalizing the abnormal vasculature in tumors, and thus improving the delivery of chemotherapeutic agents to the tumor cells. Second, chemotherapeutic drugs given in a low-dose, un-interrupted, and protracted way can induce anti-neoplasm effect through the anti-angiogenesis activity. What so-called "metronomic chemotherapy" is based on direct targeting of the activation, growth, and proliferation of vascular endothelial cells by cytotoxic chemotherapeutic agents. The anti-angiogenesis effect of metronomic chemotherapy is suppressed by VEGF/VEGFR signaling pathways and thus can be further potentiated by agents blocking those survival signals of endothelial cells. In this regard, UFUR appears to be a good candidate for metronomic chemotherapy because UFUR and its metabolites have already been shown to inhibit angiogenesis in several pre-clinical models.

The combination of tegafur/uracil (UFUR®) and thalidomide has clinical advantages for patients with HCC. Both drugs are orally active, thus are convenient to be given on an out-patient basis. More importantly, the low and non-overlapping toxicity profiles of the two drugs make the combination relatively safe in patients of HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven HCC, or HCC diagnosed by clinical criteria. The clinical diagnosis of HCC should is defined when all the following criteria are met:

   I.Chronic hepatitis B or C virus carrier; II.Presence of hepatic tumor(s) with image findings (sonography, CT scan, etc) compatible with HCC and no evidence of other gastrointestinal tumors; III.A persistent elevation of serum α-fetoprotein (AFP) level of ≧ 400 ng/ml.
2. Stage IV diseases by AJCC staging system, or loco-regional diseases which are not operable and not treatable by transarterial (chemo)embolization, percutaenous interventional therapy, or other empirical therapy of higher priority.
3. Measurable disease by RECIST criteria.
4. Karnofsky performance status ≧ 70%.
5. Age of 18 years or older.
6. Adequate liver function reserves:

   I.Class A according to Child-Pugh classification; II.Alanine aminotransferase (ALT) ≦ 5 times the ULN; III.Serum total bilirubin ≦ 1.5 times ULN.
7. Adequate bone marrow reserves:

   White blood cell (WBC) ≧ 4,000/mm3 or absolute neutrophil count (ANC) ≧ 1,500/mm3;Platelets ≧ 75,000/mm3.
8. Serum creatinine ≦ 1.5 times the ULN.
9. Previous local therapy, such as radiotherapy, hepatic arterial embolization, radiofrequency ablation, percutaenous inverventional therapy, is allowed if the treatment was completed at least 6 weeks prior to the enrollment.
10. Sexually active patients, in conjunction with their partners, must practice birth control during and for 3 months after thalidomide therapy.
11. Written informed consent.

Exclusion Criteria:

1. Concurrent radiotherapy, chemotherapy, immunotherapeutic drugs, corticosteroids or other investigational drug(s).
2. Previous exposure to the followings:

   I.Cytotoxic chemotherapy; II.Thalidomide.
3. CNS metastasis.
4. Concomitant diseases that might be aggravated by investigational drugs:

   I.Active or non-controlled infection; II.≧ NCI grade 2 peripheral neuropathy; III.History of seizures within the past 10 years or currently on anticonvulsant medication.
5. Organ transplantation.
6. Major systemic diseases those are inappropriate for systemic chemotherapy.
7. Mental status not fit for clinical trials.
8. Inability to take medications orally.
9. Pregnant or breast-feeding women.
10. Life expectancy less than 3 month.
11. Other malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ, from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Primary Objective
To assess the overall response rate of tegafur/uracil (UFUR®) and thalidomide in the treatment of advanced or metastatic hepatocellular carcinoma.

SECONDARY OUTCOMES:
Secondary Objectives
To determine the disease stabilization rate (CR+PR+SD).
To assess the progression-free survival and overall survival.
To establish the safety profile.
To evaluate the changes of circulating factors indicating the angiogenesis activity and their correlation with objective tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Huei Yeh, Ph.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Ban-Ciao, Taiwan